CLINICAL TRIAL: NCT05399940
Title: The Relationship Between Serum PSA Levels and WBC, Delta Neutrophil Index (DNI) and Other Hematological Parameters
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Ass. Prof., Hisar Intercontinental Hospital
Other Study IDs: 22/5-27
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Prostate Infection; Prostate Disease; Prostate Cancer
Keywords: prostatit
MeSH Terms: conditions — Prostatic Diseases; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: :PSA<4 ng/mL
  Interventions: Diagnostic Test: Serum PSA,Delta Neutrophil Index(DNI),WBC
- Group 2: PSA>4 ng/mL
  Interventions: Diagnostic Test: Serum PSA,Delta Neutrophil Index(DNI),WBC

INTERVENTIONS:
Diagnostic Test: Serum PSA,Delta Neutrophil Index(DNI),WBC — Urine culture, prostate volume
  Other Names: MPV,NLR,RDW

SUMMARY:
Purpose:

To find the correlation between hemogram parameters and Delta Neutrophil Index(DNI) and Serum PSA in patients presenting with the diagnosis of acute prostatitis.

Material-Metod: Serum PSA levels and hemogram parameters of patients who came to the urology outpatient clinic in January 2018 and May 2022 and were diagnosed with prostatitis were collected retrospectively.

DETAILED DESCRIPTION:
Serum PSA levels and hemogram parameters of patients who came to the urology outpatient clinic in January 2018 and May 2022 and were diagnosed with prostatitis were collected retrospectively.

WBC, neutrophil, lymphocyte, neutrophil-lymphocyte ratio, delta neutrophil index (DNI), PLT, RDW, and MPV values were determined in the Hemogram Parameters. Serum Total PSA and Free PSA values of the patients were also checked. Urine culture, urinary ultrasound, and antibiotic therapy

ELIGIBILITY:
Inclusion Criteria:

Acute prostatitis Male

-

Exclusion Criteria:

Prostate cancer Chronic prostatitis Other Urinary infections,

-

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male patients with acute prostatitis were included in the study.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Basri Cakiroglu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
re
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code